#### UNIVERSITY OF ROCHESTER MEDICAL CENTER

#### WILMOT CANCER INSTITUTE

# A patient-centered communication tool (UR-GOAL) for older patients with acute myeloid leukemia, their caregivers, and their oncologists

#### **December 17, 2021**

**Study Principal Investigator:** Kah Poh (Melissa) Loh, MBBCh BAO

Division of Hematology/Oncology University of Rochester Medical Center

James P Wilmot Cancer Center 601 Elmwood Ave, Box 704

Rochester, NY 14642

Email: Kahpoh loh@URMC.Rochester.edu

**Study Co-Investigator:** Supriya G. Mohile, MD, MS

Division of Hematology/Oncology University of Rochester Medical Center

James P Wilmot Cancer Center 601 Elmwood Ave, Box 704

Rochester, NY 14642

Email: Supriya Mohile@URMC.rochester.edu

Study Personnel: Terri Lloyd

James P Wilmot Cancer Center 601 Elmwood Ave, Box 704

Rochester, NY 14642

Phone: (585) 276-5652/ Fax: (585) 273-1042 Email: <u>Terri1 Lloyd@URMC.Rochester.edu</u>

Chandrika Sanapala

James P Wilmot Cancer Center 601 Elmwood Ave, Box 704

Rochester, NY 14642

Phone: (585) 275-4391/ Fax: (585) 273-1042

Email: Chandrika Sanapala@URMC.Rochester.edu

Jessica Bauer

James P Wilmot Cancer Center 601 Elmwood Ave, Box 704

Rochester, NY 14642

Phone: (585) 276-6562/ Fax: (585) 273-1042 Email: Jessica Bauer@URMC.Rochester.edu **Biostatisticians:** Eva Culakova, PhD

Department of Surgery
University of Rochester Medical Center

James P Wilmot Cancer Center 601 Elmwood Ave, Box 704

Rochester, NY 14642

Email: Eva Culakova@URMC.rochester.edu

# Contents

| 1.0 Background | 4 |
|--------------------------------------------------|----|
| 2.0 Aim and Hypothesis | 6 |
| 3.0. Study Design and Population | 7 |
| 4.0 Recruitment and Consent | 10 |
| 5.0 Registration | 14 |
| 6.0. UR-GOAL Intervention Tool | 16 |
| 7.0. Treatment Protocol | 19 |
| 8.0 Data Handling and Statistical Considerations | 25 |
| 9.0. Data Management | 27 |
| 10.0 Risks/Benefits | 32 |
| 11.0 Data Safety and Monitoring | 33 |
| 12.0 References | 35 |

# 1.0 Background

#### 1.1. Acute myeloid leukemia is a disease of the aging

Nearly 60% of acute myeloid leukemia (AML) diagnoses are in adults aged ≥ 60 years. For fit older patients with AML (i.e., without significant comorbidities or disabilities), the standard first-line treatment consists of intensive inpatient chemotherapy. Intensive chemotherapy provides the best chance for durable remission, but it is associated with a high treatment-related mortality (60-day mortality: 15-20%). Intensive therapy is utilized in <1% of older patients with AML seen in the community oncology setting, due to various reasons such as distance to tertiary centers and need for hospitalizations. In the last decade, low-intensity outpatient treatments (e.g., azacitidine, decitabine, venetoclax, ivosidenib, enasidenib) with reduced treatment-related mortality rates have become available. These treatments have permitted more older patients with AML, including those with comorbidities and disabilities, to receive leukemia-directed therapy. Despite these treatment options, 40-50% of diagnosed individuals do not undergo leukemia-directed therapies.

# 1.2. There is substantial heterogeneity in the health status of older patients, making treatment selection challenging

In a prospective study of 74 older patients with AML receiving intensive induction therapy, up to 69% had physical impairments, 42% had significant comorbidities, 29% had impaired cognition, and 40% were depressed. The effect these fitness-related factors have on disease progression, treatment tolerance, and response is not well understood, in part due to an underrepresentation of older patients in clinical trials. This is especially true regarding older patients with comorbidities and poor performance status. It is often challenging for oncologists to identify older patients with AML who are fit enough for intensive treatment, or fit enough to receive treatment at all. Practice patterns therefore vary.

#### 1.3. Older patients with AML often do not feel informed of their disease and treatment options.

We have previously conducted a qualitative study of 15 older patients with AML and 15 oncologists to better understand their experience during the initial AML diagnosis and treatment decision-making. Many older patients did not feel that they were adequately informed of their treatment options (Patient quote: "The only option I had was going through this. It's do or die.") Patients and oncologists perceived fitness-related factors such as physical function, comorbidities, psychological health, and cognition as important for initial treatment decision-making. Therefore, incorporating patient preferences and fitness-related factors into AML treatment decisions may facilitate communication and shared decision-making, leading to increased patient satisfaction. 15-18

#### 1.4. Best worst scaling to elicit patient preferences

Best-worst scaling (BWS) is a technique that assesses the relative importance that patients place on different aspects or attributes of care. BWS consists of choice tasks, with a minimum of three attributes (e.g., daily activities, quality of life, location of treatment, survival), in which a patient

is asked to indicate the best and worst options. The overall aim is to obtain a ranking of the attributes. This methodology is a reliable and valid technique that can help patients to consider the risks and benefits of treatment as well as to clarify and reveal their values to their oncologists, ultimately improving shared decision making. <sup>19,20</sup>

# 1.5. Information preferences vary among patients, and accurate prognostic awareness is an important component of shared decision-making.

In a multicenter prospective cohort study, we have found that older patients were less likely to prefer treatment success rates presented in percentages. We also found that over half of patients with hematologic malignancies overestimate their prognosis compared to their oncologists. Among older adults with AML, >90% thought that they could be cured, compared to 30% of oncologists. Patients with poor prognostic awareness are more likely to opt for aggressive chemotherapy<sup>23,24</sup> and less likely to utilize palliative and hospice services at the end-of-life. Older patients have lower awareness of their prognosis than younger adults. Therefore, prognostic discussion with oncologists can facilitate accurate prognostic awareness among older patients with AML (who are often incurable). We have shown that among older adults with cancer referred to geriatric oncology clinics at our center, almost 60% stated that a frank conversation about their prognosis would be helpful to them.

### 1.5. Caregivers play an essential role in decision-making

Caregivers (generally family members or friends) play an integral role in the care of older adults, <sup>30</sup>, and many assist patients with treatment decision-making and participate in prognostic discussions and. <sup>31,32</sup> Effective communication between older patients and caregivers is associated with patient and caregiver satisfaction with care, treatment adherence, and improved health outcomes. <sup>33,34</sup> In addition, clear communication between patients and caregivers can ensure that the needs of both are met. <sup>35</sup> Studies have shown that disagreements between patients and caregivers in the reporting of symptoms, description of treatment side effects and benefits, and estimates of prognosis are common. <sup>36-39</sup> Disagreement between patient and caregiver is associated with negative outcomes such as increased patient depression <sup>36</sup> as well increased caregiver anxiety, distress, depression, and burden (i.e., the latter refers to stress experienced by caregivers from providing care for patients). <sup>39-42</sup>

#### 1.6. Overall goal

Older adults with AML may benefit from help and support in understanding their treatment options. This pilot study seeks to develop and adapt a patient-centered communication tool (University of Rochester-Geriatric Oncology Assessment for acute myeloid Leukemia or UR-GOAL) and then evaluate the usability and feasibility of this tool. The UR-GOAL tool will incorporate BWS to elicit patient preferences as well as assessments of fitness and prognostic awareness. We hypothesize that this tool will be usable and feasible in this population. Once we have shown usability and feasibility, we will assess whether the UR-GOAL tool improves shared decision-making, communication, and prognostic awareness. Given that caregivers are closely involved in the care of older adults with cancer, we also seek to obtain feedback from caregivers. In addition, we will also obtain feedback from oncologists.

# 2.0 Aim and Hypothesis

## 2.1 Primary Aim

Develop and adapt a communication tool (UR-GOAL) for 10 older patients with AML.

#### 2.2 Secondary Aim

Evaluate the usability and feasibility of the UR-GOAL communication tool among 15 older patients with AML, their caregivers, and oncologists.

## 2.3 Exploratory Aim

To assess change in priorities longitudinally among 15 older patients with AML.

#### 2.4 Overall Hypothesis

The UR-GOAL will be usable and feasible.

#### 2.5 Usability and feasibility metrics

The usability and feasibility of the UR-GOAL communication tool will be evaluated based on the following:

- a) Recruitment rates (percentage of patients who are approached and agree to enroll)
- b) System Usability Scale (score on 10-item scale, ranging 0-100; higher score corresponds to greater usability)
- c) Semi-structured interviews (audio-recorded/transcribed interviews exploring perceived usefulness, barriers, and facilitators)

# 3.0. Study Design and Population

#### 3.1. Study Settings

Wilmot Cancer Institute (WCI), University of Rochester Medical Center (URMC) and its affiliated centers

### 3.2. Study Type

Aim 1: Qualitative study

Aim 2 and Exploratory Aim: Single-arm pilot study

#### 3.3. Study Population

Aim 1: We will gather feedback from 20 older patients with AML. We anticipate thematic saturation will be reached with this number of participants based on past similar research. 43,44 We will consent up to 30 patients to account for screen fail or withdrawal.

Aim 2 and Exploratory Aim: We will recruit 15 older patients with AML (and their caregivers if available) to evaluate the usability and feasibility. We will consent up to 20 patients to account for screen fail or withdrawal. We will also interview their oncologists.

#### 3.4. Inclusion and Exclusion Criteria for Patients

#### Inclusion criteria:

#### Aim 1

- Age ≥60 years (conventional definition of older age in AML)
- Established AML diagnosis (within 1 year)
- Able to provide informed consent
- English-speaking

#### Aim 2

- Age ≥60 years (conventional definition of older age in AML)
- Newly diagnosed AML
- Able to provide informed consent
- English-speaking

#### Exclusion criteria

None

#### 3.5. Inclusion and Exclusion Criteria for Caregivers (Aim 2 only)

#### Inclusion criteria:

• Selected by the patient when asked if there is a "family member, partner, friend or caregiver [age 21 or older] with whom you discuss or who can be helpful in health-related matters;" patients who cannot identify such a person ("caregiver") can be eligible for the study. A caregiver need not be someone who lives with the patient or provides

direct hands-on care. A caregiver can be any person who provides support (in any way) to the patient.

- Able to provide informed consent
- English-speaking

#### 3.6. Inclusion and Exclusion Criteria for Oncologists (Aim 2 only)

#### Inclusion criteria:

- A practicing oncologist
- At least one of their patients are recruited to the study
- English-speaking

#### Exclusion criteria

None

### 3.7. Number of Subjects

Aim 1: We plan to enroll 20 patients in 6 months. Two previous qualitative studies conducted in this population showed a recruitment of 75%-100%. Annually, from 2012-2018, WCI saw 60-70 patients aged  $\geq$ 60 years with AML.

Aim 2 and Exploratory Aim: We plan to enroll 15 patients (and their caregivers if available) in 12 months. We will be recruiting patients from WCI and WCI-affiliated sites. The WCI inpatient malignant hematology service will also be screened. We plan recruit at least 3 oncologists and up to 15 oncologists (assuming 1 patient per oncologist is enrolled).

#### 3.8. Gender of Subjects

The gender ratio of enrolled patients will be similar to that of the gender ratio of AML in older adults (approximately 1.2:1 male to female ratio).<sup>45</sup>

#### 3.9. Age of Subjects

We will recruit patients with AML aged 60 and above (from date of consent, confirmed on electronic medical record).

#### 3.10. Racial and Ethnic Origin

The Caucasian to Non-Caucasian ratio of individuals with AML is 5:1. In Rochester, New York, Whites, African Americans, and Hispanics make up approximately 65%, 30%, and 5% of the population (Race and Ethnicity in Rochester, NY statistical atlas). As enrollment is limited to English-speaking patients, we predict a higher percentage of whites. The study does not restrict enrollment based on race or ethnicity.

#### 3.11. Vulnerable Subjects

Recruitment will exclude vulnerable populations such as fetuses, neonates, children, pregnant woman, prisoners, and institutionalized individuals. We will also exclude adults who are deemed to not have decisional capacity and those who lost their consent capacity during the study period, as per their treating oncologist.

### 4.0 Recruitment and Consent

Subjects will be enrolled at the URMC WCI.

To ensure appropriate safety precautions when conducting in-person study procedures, the process for conducting in-person visits outlined in the Guidance for Human Subject Research will be followed.

### 4.1 Identification of Study Subjects, Recruitment, and Consent Procedures

Patients will be identified by treating physicians at WCI and WCI-affiliated sites, nurses of these physicians, and the study coordinator. The study coordinator will work closely with physicians and nurses to identify patients who have an established AML diagnosis (Aim 1) or have been newly diagnosed with AML (Aim 2). Given permission from the oncologist, the study team will screen clinic schedules of these oncology providers. The study coordinator will contact the physician (or designee) and inform them of patient eligibility and ask permission to approach the patient. The principal investigator will address any eligibility questions that may arise.

For **in-person consent with patients**, below are the possible scenarios for obtaining consent.

- 1. Physician/Study Investigator makes the initial contact and provides consent form, and patient signs consent with the physician on the same day: After confirming with the physician (or their designee) that a patient is a potential candidate for the study, the study staff will provide a consent form to the treating physician/study investigator so he/she can provide it to the patient during an in-person clinic visit. The physician/study investigator will go over every detail of the study during the clinic visit with patient. If agrees, the patient will sign the consent form with the physician/study investigator during the same in-person visit.
- 2. Study staff makes the initial contact and provides consent form, and patient signs consent with the study staff on the same day: After confirming with the physician (or their designee) that a patient is a potential candidate for the study, the patient will be provided with an informed consent form by the study staff when they come in for an inperson clinic visit. The study staff will introduce the study to the patients and go over every detail of the study. If agrees, the patient will sign the consent form with the study staff during the same in- person visit with the study staff.

For **verbal consent with patients**, below are the possible scenarios for obtaining consent.

1. <u>Physician/Study Investigator makes the initial contact, study staff follows up with the patient on the phone, and patient provides verbal consent on the phone is a patient provided to the patient on the phone is a patient provided to the patient of the pati</u>

the phone: After confirming with the physician (or their designee) that a patient is a potential candidate for the study, the physician/study investigator confirms with the patient that he/she is willing to speak with the study staff about the study. The study staff will then call the patient via phone. The study coordinator will use the verbal consent script as a written aid and will go over every detail of the study with the patient to recruit them for the study. Study staff will sign and date it to confirm that he/she followed the script and the patient agrees to participate in the study. An information sheet summarizing the study and patient's involvement will be mailed /emailed to the patient for their records.

- 2. Physician/Study Investigator makes the initial contact and provides consent form, study staff follows up with the patient on the phone, and patient provides verbal consent on the phone: After confirming with the physician (or their designee) that a patient is a potential candidate for the study, the study staff will provide a consent form to the treating physician/study investigator so he/she can provide it to the patient during an in-person clinic visit. If the patient is interested but does not want to consent on the same day, the patient will bring the consent form home. The study staff will then call the patient via phone. The study coordinator will use the verbal consent script as a written aid and will go over every detail of the study with the patient to recruit them for the study. Study staff will sign and date it to confirm that he/she followed the script and the patient agrees to participate in the study. An information sheet summarizing the study and patient's involvement will be mailed/emailed to the patient for their records.
- 3. Study staff makes the initial contact and provides consent form, study staff follows up with the patient on the phone, and patient provides verbal consent on the phone: After confirming with the physician (or their designee) that a patient is willing to speak with the study coordinator about the study, the patient will be provided with an informed consent form by the study staff when they come in for an inperson clinic visit. If the patient is interested but does not want to consent on the same day, the patient will bring the consent form home. The study staff will then call the patient via phone. The study coordinator will use the verbal consent script as a written aid and will go over every detail of the study with the patient to recruit them for the study. Study staff will sign and date it to confirm that he/she followed the script and the patient agrees to participate in the study. An information sheet summarizing the study and patient's involvement will be mailed/emailed to the patient for their records.

For caregivers, we will obtain verbal consent. They will be provided with an information sheet. The patient will identify a caregiver and makes the initial contact. After confirming with the

patient that a caregiver is willing to speak with the study coordinator about the study, the study staff then call the caregiver via phone. The study coordinator will use the verbal consent script as a written aid and will go over every detail of the study with the caregiver to recruit them for the study. Study staff will sign and date it to confirm that he/she followed the script and the patient agrees to participate in the study. An information sheet summarizing the study and caregiver's involvement will be provided/mailed/emailed to the caregiver for their records.

For oncologists, we will obtain verbal consent and they will be provided with an information sheet.

#### 4.1.1. Informed Consent

Informed consent will be obtained from the patient by the study investigators or coordinators. Consent documents will be signed by the patient and maintained in the patient record with copies provided to the patient. For verbal consent, documents will be maintained in the patient record with copies provided to the patient. Verbal consent documents with caregivers and oncologists will also be maintained in separate records with copies provided to caregivers and oncologists.

#### Waiver of documentation of consent:

We are requesting for waiver of documentation of consent as the research involves no more than minimal risk to the subjects and involves procedures for which written consent is normally not required outside the research context. The only record linking the subject and the research would be the consent document and the principal risk would be potential harm resulting from a breach of confidentiality.

#### Alteration of HIPAA Authorization:

We are requesting an alteration of HIPAA authorization. We will provide an information sheet to patients who provided verbal consent. Verbal consent will allow for reduction of in-person visits, thus maximizing the safety of both patients and study staff. Nonetheless, when possible and if we are able to coordinate study and clinic visits, we will obtain written informed consent.

The study cannot be conducted without the use of protected health information (PHI) as we have to link patient reported data with medical history collected on electronic medical record. We have adequate plans to protect the PHI from improper use and disclosure. We will destroy identifiers after completion of the study for 7 years. We will not reuse or disclose the PHI to another person or entity other than the study investigators. The waiver will not adversely affect the privacy rights of the individual and the research cannot be practicably done without access to the use of the PHI.

We are requesting an alteration of HIPAA authorization for enrollment of caregivers and oncologists. We will provide an information sheet to these participants who provided verbal consent. Verbal consent will allow for reduction of in-person visits, thus maximizing the safety of both patients and study staff. We are not collecting protected health information (PHI) from Oncologists or Caregivers.

### 4.1.2. Human Subject Protection

The University of Rochester Research Subject Review Board Investigator Guidance policy will be used to ensure that ethical standards for human subjects are upheld.

#### 4.1.3. Participation

Regulations at the state, federal, and institutional level will be adhered to in regards to informed consent. Study participation is completely voluntary. After consenting, participants may withdraw from the study at any time for any reason, and they may do so without any repercussions. Participants may also be withdrawn by study personnel if it is determined that it is not favorable for the patient. All information regarding consent and withdrawal will be kept confidential.

#### 4.1.4. Duration

Aim 1: The qualitative section of this study involves interviewing consented patients for 30-60 minutes. They will watch an education video and use the UR-GOAL tool and feedback can be provided during the interview. Study participants will be interviewed by the study team either in-person (in a private space) or via phone/zoom. Interviews will be audio-recorded, uploaded to Box, and subsequently deleted from the audio-recorder.

Aim 2 and Exploratory Aim: After completing baseline measures, watching an education video, and completing the UR-GOAL tool, study participants will participate in a semi-structured interview with the study team for 30-60 minutes either in-person or via phone/zoom. The post-intervention measures will be completed within 1-2 weeks of the patient's encounter with the primary oncologist either in-person or via phone/zoom. Caregivers will complete baseline measures and watch an education video. They will participate in a separate semi-structured interview with the study team for 30-60 minutes either in-person or via phone/zoom. The post-intervention measures will be completed within 1-2 weeks of the patient's encounter with the primary oncologist either in-person or via phone/zoom. After the study is completed, participant data will be maintained for 7 years at URMC and will be kept in a password-protected database.

Oncologist will also complete the post-intervention assessments (surveys) within 1-2 weeks of the patients encounter. Oncologists will participate in a semi-structured interview with the study team for 30-60 minutes either in-person or via phone/zoom., after at least one of their patients have completed the tool. The semi-structured interviews with oncologists will be conducted at any time during the study. After the study is completed, participant data will be maintained for 7 years at URMC and will be kept in a password-protected database.

# 5.0 Registration

If patients, caregivers, and oncologists meet eligibility criteria and have provided informed consent, the study personnel will enter the following information into the OnCore Database:

#### 5.1. Registration Information for Patients

- 5.1.1 Site
- 5.1.2 Most recent IRB approval date
- 5.1.3 Name of person registering study participant
- 5.1.4 Eligibility verification
- 5.1.5 Verification that consent form has been signed and who signed by (patient and/or health care proxy) and date signed
- 5.1.6 Treatment facility (WCI vs. Other)
- 5.1.7 Participant's identification
  - 5.1.7.a First and last names
  - 5.1.7.b Birth date (MM/DD/YEAR)
  - 5.1.7.c Gender
  - 5.1.7.d Race
  - 5.1.7.e Five-digit zip code
  - 5.1.7.f Medical Record Number
  - 5.1.7.g Ethnicity
  - 5.1.7.h Patient's preferred and alternate phone numbers (and email address if patients consent to be contacted via email)
  - 5.1.7.i Date of baseline visit

#### 5.2. Registration Information for Caregivers

- 5.2.1 Participant's identification
  - 5.2.1.a First and last names
  - 5.2.1.b Birth date (MM/DD/YEAR)
  - 5.2.1.c Gender
  - 5.2.1.d Race
  - 5.2.1.e Five-digit zip code
  - 5.2.1.f Ethnicity
  - 5.2.1.g Caregiver's preferred and alternate phone numbers (and email address if patients consent to be contacted via email)

#### 5.3. Registration Information for Oncologists

- 5.3.1 Participant's identification
  - 5.3.1.a First and last names
  - 5.3.1.b Birth date (MM/DD/YEAR)
  - 5.3.1.c Gender
  - 5.3.1.d Race
  - 5.3.1.e Five-digit zip code
  - 5.3.1.f Ethnicity

## 5.4. Initial Assessment

In Aim 1, study patients will complete demographics and a 30-60 minutes interview in which they will watch an education video and complete the UR-GOAL tool and provide feedback. Patients in Aim 2 will complete baseline assessments with the study coordinator, watch an education video, and complete the UR-GOAL tool. Caregivers in Aim 2 will complete baseline assessments with the study coordinator and watch an education video.

#### 6.0. UR-GOAL Intervention Tool

The proposed tool consists of three components: BWS to elicit patient preferences, fitness assessment, and prognostic awareness assessment (Figure 1). In addition, an education video will also be included. The education tool provides information on the diagnosis, epidemiology, symptoms, risk factors, and prognosis of AML, as well as goals of AML treatment and treatment approaches.

Figure 1: Components of the UR-GOAL communication tool



#### 6.1.Best-worst scaling

BWS consists of 10 choice tasks, with 4 attributes per task. Patients will be presented with 4 attributes at a time, in which a patient is asked to rank the most and least important attribute when choosing a treatment (**Figure 2**). This process then repeats 10 times until all attributes are evaluated. Based on our qualitative study of older patients with AML and oncologists, <sup>43</sup> we selected eight attributes that are important in treatment decision making. At completion, a summary containing the ranking of the attributes will be provided to the patient and oncologist. The patient summary also includes a question prompt list (based on their top four attributes).

Figure 2: Best-Worst Scaling showing 4 options

Please consider how important the priorities below are to you when choosing a cancer treatment. Considering only these 4 priorities, what is the MOST IMPORTANT and which is the LEAST IMPORTANT?

| Daily activities Whether or not I will be able to do the activities that I do now without help Quality of life How likely it is that my quality of life will change Location of treatment Whether a treatment requires a one-month stay at the hospital versus receiving it in the hospital and going home on the same day Survival How likely it is that I will be alive one year after treatment | wost imp | Urtant | east important |
|---|---|---|---|
| Quality of life How likely it is that my quality of life will change Location of treatment Whether a treatment requires a one-month stay at the hospital versus receiving it in the hospital and going home on the same day Survival | $\bigcirc$ | Daily activities | $\bigcirc$ |
| How likely it is that my quality of life will change Location of treatment Whether a treatment requires a one-month stay at the hospital versus receiving it in the hospital and going home on the same day Survival | | Whether or not I will be able to do the activities that I do now without | help |
| Location of treatment Whether a treatment requires a one-month stay at the hospital versus receiving it in the hospital and going home on the same day Survival | $\bigcirc$ | Quality of life | $\circ$ |
| Whether a treatment requires a one-month stay at the hospital versus receiving it in the hospital and going home on the same day Survival | | How likely it is that my quality of life will change | |
| receiving it in the hospital and going home on the same day Survival | | Location of treatment | |
| | | · | rsus |
| How likely it is that I will be alive one year after treatment | $\bigcirc$ | | $\bigcirc$ |
| | | How likely it is that I will be alive one year after treatment | |

#### 6.2. Fitness Assessment:

We will include assessments (e.g., physical function, nutritional status; Table 1) that evaluate fitness and are important in decision-making for both patient and oncologist.<sup>13</sup> At completion, a summary containing the patient's fitness level will be provided to the oncologists.

Table 1: Questionnaires that will be included in the tool

| Fitness domain | Assessments |
|---|---|
| Physical function | Activities of daily living, instrumental |
| | activities of daily living, number of falls, |
| | Short Physical Performance Battery |
| Nutritional status | Weight loss in the prior 6 months |
| Comorbidity | Hearing and eyesight |
| Psychological health | Geriatric Depression scale |
| Social support | Patient's social support |
| | Living situation |
| Medications | Number of medications |
| Cognition | Mini-Cog |

#### 6.3. Prognostic Awareness Assessment:

We will incorporate assessment of prognostic awareness (i.e., chance of cure and survival estimates, their information preference (i.e., do they prefer treatment success rate presented in percentages, words, fractions, or they wanted to hear about a previous patient that the physician treated), and whether conversation about prognosis would be helpful to them. At completion, a summary contacting this information will be provided to the oncologists.

As described above, the generated summaries are tailored and intended to improve communication between the patient and oncologist during the decision-making process.

#### 6.4. Education Video

As the overall goal of the study is to improve patient-physician communication, we created an education video for patients. The video contains basic information about the diagnosis, epidemiology, symptoms, risk factors, and prognosis of AML, as well as goals of AML treatment and treatment approaches. We created this video because of two main reasons: 1) Our preliminary data suggest that many older patients may not understand the AML diagnosis and treatment approaches given the acuity, 2) The video provides an overview of AML which will help patients complete the tool subsequently (e.g., the tool will ask patients if they are willing trade quality of life for higher remission, and the education video provides information on what remission means in the context of the different treatments). The video is not part of standard of care. We developed this video based on feedback from the leukemia and bone marrow transplant and geriatric oncology groups at WCI.

The video is available for view using this link: <a href="https://rochester.box.com/s/m25aidirevgzaeumgvnpxmd3mck1lxhy">https://rochester.box.com/s/m25aidirevgzaeumgvnpxmd3mck1lxhy</a>

#### 7.0. Treatment Protocol

#### 7.1. Study Outline

We will screen and consent eligible patients of treating physicians at WCI and WCI-affiliated centers.

For Aim 1, the study team will conduct an in-person or zoom/phone interview for 30-60 minutes. First, we will explain the rationale of the study. Second, patients will use the communication tool. Third, we will conduct an interview to elicit feedback about the communication tool. This feedback will be used to adapt the tool for Aim 2.

For Aim 2 and Exploratory Aim (Figure 3), the study subject will complete baseline measures and utilize the UR-GOAL communication tool either in-person or via zoom/phone. Following this, patients will complete the usability testing form. The patient (and caregiver if available) will have a visit with their primary oncologist and the clinical encounter will be audio-recorded. The study staff will provide an audio recorder to the physician for in-person or phone visits, and the zoom recording feature will be used for zoom visits. All parties present for recorded visits, including: enrolled patients, any accompanying caregivers, family or friends, the oncologist, and any other physicians or health care providers not participating in the study will be fully aware that the conversation is being audio-recorded before any recording begins, in addition to the prior written consent of enrolled patients. Patients, caregivers and oncology physicians may receive copies of these recordings at their request.

The post-intervention measures, including the qualitative interviews, for patients and caregivers will be completed within 1-2 weeks of the patient's encounter with the primary oncologist either in-person or via phone/zoom. The interviews will be conducted separately. Patients will participate in a semi-structured interview for 30-60 minutes during which feedback will be elicited. Enrolled caregivers will also participate in a separate semi-structured interview for 30-60 minutes during which feedback will be elicited. Oncologist will also complete the post-intervention assessments (surveys) within 1-2 weeks of the patients encounter. The semi-structured interviews with oncologists will be conducted at any time during the study, after at least one of their patients have completed the study procedures.

To assess priorities longitudinally, patients will complete the BWS on the tool at 1, 2, 3, and 6 months.

Figure 3: Study Procedures (Aim 2 and Exploratory Aim)



### 7.2. Assessments of the Participants

Demographic, clinical, and cancer characteristics will be collected.

#### 7.2.1. Demographics – Patient, Caregiver, and Oncologist

Patient and caregiver's age, date of birth, race, ethnicity, gender, highest level of education achieved, employment status, and marital status. This will only be collected at baseline.

Oncologist's name, date of birth, race, five-digit zip code, ethnicity, and gender will be collected.

#### 7.2.2. Clinical and Cancer Characteristics - Patient

ECOG performance status, diagnosis, prior hematologic malignancies, cytogenetic risk group and treatment regimen will be abstracted from the medical records. This information will only be collected at baseline.

#### 7.2.3. Measures

Measures will be collected via the UR-GOAL tool, done in person, or mailed to the participants.

#### 7.2.2.1. Physical Function and Functional Status (Baseline Only - Patient)

Short Physical Performance Battery (SPPB; baseline only): The SPPB is an objective physical assessment evaluating lower extremity physical function. It is comprised of a four-meter walk, repeated chair stands and a balance test. Impairment on SPPB testing has been shown to be predictive of short-term mortality and nursing home admission in community-dwelling older adults.<sup>46</sup> If in-person SPPB cannot be performed, we will

perform the virtual SPPB via the phone/zoom, which evaluates the participants' perceived ability to perform above tests (walking, repeated chair stands, and balance).<sup>47</sup>

Activities of daily living (ADL): ADLs are measures of self-care. ADL independence will be assessed using the Katz Index of Independence in Activities of Daily Living, commonly referred to as the Katz ADL. The Katz ADL is the most appropriate instrument to assess functional status as a measurement of the client's ability to perform activities of daily living independently. Clinicians typically use the tool to detect problems in performing activities of daily living and to plan care accordingly. The Index ranks adequacy of performance in the six functions of bathing, dressing, toileting, transferring, continence, and feeding. Clients are scored yes/no for independence in each of the six functions. A score of 6 indicates full function, 4 indicates moderate impairment, and 2 or less indicates severe functional impairment.<sup>48</sup>

*Instrumental Activities of Daily Living (IADL):* Self-reported functional status will be assessed using the IADL subscale of the Multidimensional Functional Assessment Questionnaire: Older American Resources and Services (OARS). The IADL subscale consists of seven questions rated on a three-point Likert scale. It measures the degree to which an activity can be performed independently.<sup>49</sup>

*Fall History:* A self-reported history of falls in the past three months will be recorded. A history of a recent fall has been demonstrated to be independently predictive of increased risk for chemotherapy toxicity in older cancer patients.<sup>50</sup>

#### 7.2.2.2. Nutritional Status (Baseline Only - Patient)

Screenings for nutritional deficit will be performed with body mass index (BMI) evaluation and self-reported weight loss.

#### 7.2.2.3. Comorbidity (Baseline Only - Patient and Caregiver)

*OARS Comorbidity:* Patients and caregivers report coexisting illnesses and indicate the degree to which these comorbidities interfere with their daily activities.<sup>51</sup>

Patients and caregivers also self-report their perceived levels of eyesight and hearing.

#### 7.2.2.4. Psychological Health (Baseline and Post-Intervention – Patient and Caregiver)

General Anxiety Disorder-7: A 7-item screening tool for anxiety.<sup>52</sup>

*Geriatric Depression Scale-15:* A 15-item valid and reliable screening tool for depression in older adults.<sup>53</sup> This will be used for patients.

*Patient Health Questionnaire-2 (PHQ-2)*: A 2-item valid and reliable screening tool depression in the general population.<sup>54</sup> This will be used for caregivers.

#### 7.2.2.5. Social Support (Baseline Only - Patient)

*OARS Medical Social Support:* A 13-item questionnaire for patients regarding persons involved in medical social support as well as perception of overall support. 51,55

Patients also self-report their living situation and their main social support.

### 7.2.2.6. Medications (Baseline Only - Patient)

*Medications:* We will record all prescription and non-prescription medications, dosage and frequencies from the medical records. Polypharmacy is defined as the use of 5 or more medications.

#### 7.2.2.7. Cognition (Baseline Only - Patient)

*Mini-Cog (baseline only):* A 3-item screening tool for cognitive impairment in older adults.<sup>56</sup>

# <u>7.2.2.8. Communication Self-Efficacy (Baseline and Post-intervention – Patient and Caregiver)</u>

*Perceived Efficacy in Patient-Physician Interactions (PEPPI):* A valid and reliable assessment of perceived self-efficacy of older patients interacting with physicians.<sup>57</sup>

Perceived Efficacy in Caregiver-Physician Interactions (PECPI): A valid and reliable assessment of perceived self-efficacy of caregivers interacting with physicians.<sup>58</sup>

# <u>7.2.2.9. Patient-Centered Communication (Post-Intervention Only – Patient and Caregiver)</u>

Patient-Centered Communication in Cancer Care (PCC-Ca-36): A questionnaire assessing patient-centered communication in six domains: exchanging information, making decisions, fostering healing relationships, enabling patient self-management, managing uncertainty, and responding to emotions. <sup>59</sup>We will adapt the PCC-Ca-6 for caregivers.

# 7.2.2.10. Shared Decision-Making (Post-Intervention Only – Patient, Caregiver, and Physician)

*Shared Decision-Making Questionnaire (SDM-Q-9):* A 9-item reliable questionnaire assessing patient satisfaction with the medical decision-making process.<sup>60</sup>

Shared Decision-Making Questionnaire (SDM-Q-Doc): A 9-item reliable questionnaire assessing physician satisfaction with the medical decision-making process.<sup>61</sup>

CollaboRATE Measure: A 3-item questionnaire assessing patient, caregiver, and

physician shared decision-making.<sup>62</sup>

Preparation for Decision Making Scale: A 10-item questionnaire assessing patients' and caregivers' perception of how useful the communication tool is in preparing them to communicate with their physician at a consultation focused on making a health decision.<sup>63</sup>

#### 7.2.2.11. Disease Knowledge (Baseline and Post-intervention – Patient and Caregiver)

*Disease Knowledge*: A 14-item questionnaire assessing patients and caregivers' understanding of AML.

# 7.2.2.12. Information and Decision-Making Preferences (Baseline Only – Patient and Caregiver)

*Information Preferences:* A questionnaire assessing patient and caregiver preferences regarding treatment information.

*Decision-Making Preferences:* The Control Preference Scale assess patient and caregivers' preferred roles in treatment decisions.<sup>64</sup>

#### 7.2.2.13. Disease Understanding (Patient, Caregiver, and Physician)

Disease Understanding – Patient (baseline and post-intervention): A questionnaire assessing patient's prognostic understanding of illness and preferences regarding life expectancy discussions.

Disease Understanding – Caregiver (baseline and post-intervention): A questionnaire assessing caregiver's prognostic understanding of illness and preferences regarding life expectancy discussions.

Disease Understanding – Physician (post-intervention only): A physician-facing questionnaire assessing patient prognosis.

# 7.2.2.14 Decisional conflict and regret (post-intervention for decisional conflict and 1, 2, 3, and 6 month for decisional regret at)

*Decisional conflict scale* – A questionnaires that measures personal perceptions of uncertainty in choosing options, modifiable factors contributing to uncertainty, and effective decision making.<sup>65</sup>

*Decisional regret scale* – A questionnaire that measures distress or remorse after a healthcare decision.<sup>66</sup>

Was it worth it questionnaire – A questionnaires that assesses satisfaction with decision made <sup>67</sup>

#### 7.2.2.15 Health-related quality of life (Post-Intervention and 1, 2, 3, and 6 month)

EQ-5D-5L: A health-related quality of life questionnaire that consists of five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.<sup>68</sup>

## 7.2.2.16. Usability (Post-Intervention Only)

*Usability questions – Patient and Oncologist*: Questions to assess usability of the tool and/or summary.

### 7.2.2.17. Environmental Mastery (Baseline and Post-Intervention - Caregiver)

*Ryff's Environmental Mastery:* A 7-item questionnaire measuring whether the respondent makes effective use of opportunities and has a sense of mastery in managing environmental factors and activities, including managing everyday affairs and creating situations to benefit personal needs.<sup>70</sup>

# 8.0 Data Handling and Statistical Considerations

## 8.1. Data Handling

<u>8.1.1.</u> The same protocols and procedures for data quality and control that are readily used for the NCI Community Oncology Research Program (NCORP) Research Base protocols currently being overseen by our office (which have accrued over 1,000 patients in the previous year) will be used for this study. Patients will fill out forms generated from RedCap and this information will be entered into RedCap (Section 9.5). Study personnel will perform SPPB and the scores will be entered into RedCap.

8.1.2. It is anticipated that allowing for the appropriate number of evaluable participants and by checking self-report measures for completeness, we will have a full complement of data. Every effort will be made to encourage and facilitate participants' completion of all questionnaires and all items on the questionnaires for each study assessment. In the event that missing data occur, every effort will be made to contact participants via phone and obtain the data or to find out why the questionnaires or items are missing. The reasons for missing data will be documented. Missing questionnaire items will be treated in accordance with the documented scoring procedures. Although it is very unlikely that missing values will not occur randomly, we will confirm their randomness. Multiple imputation<sup>71</sup> will be applied to (1) give more accurate statistical tests and standard errors for key treatment effect parameters and to (2) give some indication of the sensitivity of the analyses to missing data. The causes and pattern of the missing data will be examined and taken into consideration in the design of future studies.

8.1.3. Data collected via the UR-GOAL communication tool will only be accessed by the following: 1) The research team and 2) The treating physician and their designee.

## 8.2. Data Analysis and Sample Size:

#### 8.2.1. Analysis Plan for Aim 1

We anticipate thematic saturation will be reached with this number of participants (N=20) based on past similar research. 43,44 We will conduct and audio-record all interviews, which will be transcribed by a professional transcription service. We will analyze the qualitative data using grounded theory and constant comparative methods, with coding to structure data into categories and create groups according to the broader issues or themes. 72 An audit trail of the coding activity will be kept. We will critically examine the data collection and analysis process and reach consensus on key themes from patient feedback to be used to adapt the intervention in preparation for Aim 2.

#### 8.2.2. Analysis Plan for Aim 2

We anticipate that our proposed sample size will be sufficient based on prior research<sup>73</sup> and also published guidance on usability study.<sup>74,75</sup> The feasibility of the UR-GOAL tool

will be evaluated based on the percentage of patients consented to the study ultimately completing all study components.

Recruitment rate (percentage of patients who are approached and agree to enroll) will also be described. Other feasibility metrics include retention rate (percentage of patients who were enrolled and completed the intervention and assessments). The usability of the UR-GOAL tool will be evaluated using the SUS score.

We will consider the UR-GOAL study feasible if >50% of consented patients ultimately complete all study components. We chose 50% based on our prior behavioral intervention study in this population and published studies that utilize similar tools (e.g., value elicitation tool). <sup>73,76,77</sup> We will use descriptive statistics to describe the measures. If we do not meet our usability and feasibility goals, we will further adapt the study and tool.

For other measures, these are being collected in preparation for a larger clinical trial in the future. As exploratory analyses, paired t-tests or McNemar's test will be used to evaluate change in measures from baseline to post-intervention. Linear mixed models will be used to assess change in measures over several time points.

Qualitative data from the semi-structured interviews will be analyzed as per Aim 1. Interviews will be conducted, audio-recorded, and transcribed. We will analyze the qualitative data using grounded theory and constant comparative methods, with coding to structure data into categories and create groups according to the broader issues or themes.<sup>72</sup> An audit trail of the coding activity will be kept. We will critically examine the data collection and analysis process and reach consensus on key themes from patient feedback to be used to further adapt the tool.

For audio-recorded clinic encounters, we will use published shared decision-making coding schemes to assess quality of shared decision making. <sup>78,79</sup> Coders will undergo extensive training and supervision by study investigators.

# 9.0. Data Management

# 9.1. Data Collection Table

# 9.1.1. Aim 1

| 7.1.1. Allii I | Eligibility<br>and Consent<br>Form | Assessment |
|---|---|---|
| Informed Consent | X | |
| Demographics | | X |
| Clinical and Cancer Characteristics | | X |
| Qualitative Interview | | X |
| Short Physical Performance Battery/Virtual Short Physical Performance Battery, Activities of Daily Living, Instrumental Activities of Daily Living, Fall History | | X |
| Nutritional Status | | X |
| Comorbidity | | X |
| Geriatric Depression Scale-15 (GDS-15),<br>Generalized Anxiety Disorder-7 (GAD-7) | | X |
| Social Support | | X |
| Medications | | X |
| Mini-Cog | | X |
| Information and Decision-Making Preferences | | X |
| Disease Understanding - Patient | | X |

# 9.1.2. Aim 2 a) Patients

| | SCHEDULE OF DATA COLLECTION | | | |
|---|---|---|---|---|
| | Eligibility and<br>Consent Form | Baseline<br>Assessment<br>(week 0) | Post-intervention<br>Assessment (week 1-<br>2) | Month 1, 2, 3, and 6 |
| Informed Consent | X | | | |
| Demographics | | X | | |
| Clinical and Cancer Characteristics | | X | | |
| Qualitative Interview | | | X | |
| Short Physical Performance Battery/Virtual Short Physical Performance Battery, Activities of Daily Living, Instrumental Activities of Daily Living, Fall History | | X | | |
| Nutritional Status | | X | | |
| Comorbidity | | X | | |
| Geriatric Depression Scale-15<br>(GDS-15),<br>Generalized Anxiety Disorder-7<br>(GAD-7) | | X | X | |
| Social Support | | X | | |
| Medications | | X | | |
| Mini-Cog | | X | | |
| Perceived Efficacy in Patient-<br>Physician Interactions (PEPPI) | | X | X | |
| Patient-Centered Communication in Cancer Care (PCC-Ca-36) | | | X | |
| Shared Decision-Making (SDM-Q-9) <sup>a</sup> | | | X | |
| CollaboRATE Measure | | | X | |
| Preparation for Decision Making<br>Scale | | | X | |
| Patient Disease Knowledge | | X | X | |
| Information and Decision-Making<br>Preferences - Patient | | X | | |
| Disease Understanding - Patient | | X | X | |
| Decisional Conflict Scale Decisional Regret Scale and Was it Worth It Questionnaire | | | X | X |
| BWS component only of the tool | | | | X |
| EQ-5D-5L | | | X | X |
| Usability (Usability questions) | | | X | |

b) Caregivers

| | SCHEDULE OF DATA COLLECTION | | |
|---|---|---|---|
| | Eligibility<br>and Consent<br>Form | Baseline<br>Assessment<br>(week 0) | Post-<br>intervention<br>Assessment<br>(week 1-2) |
| Informed Consent | X | | |
| Demographics | | X | |
| Qualitative Interview | | | X |
| Comorbidity | | X | |
| Patient Health Questionnaire-2 (PHQ-2),<br>Generalized Anxiety Disorder-7 (GAD-7) | | X | X |
| Perceived Efficacy in Caregiver-Physician Interactions (PECPI) | | X | X |
| Patient-Centered Communication in Cancer Care (PCC-Ca-6) – adapted caregiver version | | | X |
| Ryff's Environmental Mastery | | X | X |
| CollaboRATE Measure | | | X |
| Preparation for Decision Making Scale | | | X |
| Caregiver Disease Knowledge | | X | X |
| Information and Decision-Making Preferences – Caregiver | | X | |
| Disease Understanding – Caregiver | | X | X |

c) Oncologists

| | SCHEDULE OF DATA COLLECTION | | |
|---|---|---|---|
| | Eligibility<br>and Consent<br>Form | Baseline<br>Assessment<br>(week 0) | Post-intervention<br>Assessment (week<br>1-2) |
| Informed Consent | X | | |
| Demographics | | X | |
| Shared Decision-Making (SQM-Q-Doc, physician version) | | | X |
| Disease Understanding – Physician | | | X |

| Usability questions | X |
|---|---|
| Qualitative Interview | After at least 1 patient per oncologist completed study procedures, can be done at any point during the study |

- 9.2. All hardcopy research records will be stored onsite in the URMC, in locked research files at the WCI. The Cancer Center is secured with electronic key cards. Offices within the Cancer Center are again secured by key and data is kept in locked file cabinets. Electronic research records are stored on the URMC's password secured and firewall protected networks. These are the same methods of security used for patient medical records. For audio-recordings, these will be uploaded to Box within a week of the interview and deleted from the audio-recorded. All study data will be kept for a period of 7 years after the study and all reports and publications are complete.
- 9.3. All data collected for the current study will be used in post hoc analyses as appropriate. Data will not be used for future studies without prior consent of the patient. The patient's individual research record will not be shared with their treating physician, unless they provide consent or the patient's treating physician is a study physician, in which case they will have access to study data as a study co-investigator. Overall study results will be presented to participants, faculty and staff at the URMC after completion of the study. Study results will be presented at professional meetings and published.
- 9.4. The study coordinator will assign a numerical study ID to each participant once they have signed the consent form (chronologically based on the data they signed consent i.e., 001, 002, 003...). All study forms and questionnaires will use this number and the participant's first, middle, and last initials as identifiers, to ensure data integrity. Other identifying information will not exist on these forms. A complete list of study participants with study ID, name, and contact information will be maintained separately. This linkage information will only be accessible to the study coordinator, study investigators, and the individuals responsible for maintaining the database.
- 9.5. Additionally, data on the socio-demographics, clinical, and cancer and treatment characteristics will be collected and managed by the research teams at URMC using REDCap electronic data capture tools hosted at URMC.<sup>80</sup> We will also evaluate the medical records for clinical characteristics and outcomes, and utilize REDCap to collect and manage this information.
  - 9.5a. URMC provides the following information on the **REDCap program:** "Vanderbilt University, in collaboration with a consortium of institutional partners, has developed a software toolset and workflow methodology for electronic collection and management of research and clinical trial data, called REDCap (Research Electronic Data Capture). The REDCap system is a secure, web-based application that is flexible enough to be used for a

variety of types of research. It provides an intuitive interface for users to enter data and real time validation rules (with automated data type and range checks) at the time of data entry. REDCap offers easy data manipulation with audit trails and functionality for reporting, monitoring and querying patient records, as well as an automated export mechanism to common statistical packages (SPSS, SAS, Stata, R/S-Plus). Through the REDCap Consortium, Vanderbilt has disseminated REDCap for use around the world. Currently, over 240 academic and non-profit consortium partners on six continents with over 26,000 research end-users use REDCap.<sup>81</sup>

- **9.5b.** According to the Clinical and Translational Science Institute (CTSI), REDCap is supported with the following means. "The CTSI Informatics Core, a unit of the SMD Academic Information Technology (AIT) Group, will serve as a central facilitator for data processing and management. REDCap data collection projects rely on a thorough study-specific data dictionary defined in an iterative self-documenting process by all members of the research team, with planning assistance from the AIT-CTSI Informatics Core. The iterative development and testing process results in a well-planned data collection strategy for individual studies."<sup>72</sup>
- **9.5c.** The CTSI states that regarding security, "REDCap servers are housed in a local data center at the University of Rochester and all web-based information transmission is encrypted. REDCap was developed in a manner consistent with HIPAA security requirements and is recommended to University of Rochester researchers by the URMC Research Privacy Officer and Office for Human Subject Protection. 81

## 10.0 Risks/Benefits

#### 10.1. Risks

There is potential loss of confidentially associated with participation in the proposed study. In terms of loss of confidentiality, quantitative data from participants will need to be stored. Though rigorous and well-tested data safety and security guidelines will be observed, there is still a chance that confidentiality could be breached and sensitive medical information could become known to persons outside the research team.

#### 10.2. Benefits

There are no anticipated benefits to the participants.

#### 10.3 Payments and Costs

Patients participating in the first aim will be paid \$30 and those participating in the second aim will be paid \$50 for their participation in the form of gift cards. For Aim 1, participants will receive the gift cards immediately following the interviews. For Aim 2, participants will be paid for completion of the post-intervention assessment. Oncologists will not be reimbursed for their participation.

# 11.0 Data Safety and Monitoring

Only adverse events (AEs) related to the study intervention or procedures will be reported. In other words, AEs related to cancer treatment will not be reported.

#### 11.1. Adverse Event Reporting Requirements

<u>11.1.1.</u> Adverse events will be reported using the URCC Adverse Event form and/or as required by the Cancer Center Clinical Trials Office.

| | Grade 1 | Grade 2 | | | | Grade 3 | | | Grade 4 | | Grade 5 | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| | | Unexpe | ected | Expected Unexpected Expected Unexpected Expected | | Unexpected | | Unexpected Expected | | Expected | Unexpected | Expected |
| | Unexpected<br>and Expected | with<br>hospitalizatio<br>n | without<br>hospital-<br>ization | | with<br>hospitalizati<br>on | without<br>hospitaliza<br>tion | with<br>hospitaliz<br>ation | without<br>hospitaliz<br>ation | | | | |
| Unrelated<br>Unlikely | Not<br>Required | Not<br>Required | Not<br>Required | Not<br>Required | Not<br>Required | Not<br>Required | Not<br>Required | Not<br>Required | 10<br>Calendar<br>Days | Not<br>Required | 10<br>Calendar<br>Days | 10<br>Calendar<br>Days |
| Possible<br>Probable<br>Definite | Not<br>Required | 10 Calendar<br>Days | Not<br>Required | Not<br>Required | 10 Calendar<br>Days | 10<br>Calendar<br>Days | Not<br>Required | Not<br>Required | 5 Calendar<br>Days | 10<br>Calendar<br>Days | 5 Calendar<br>Days | 10<br>Calendar<br>Days |
| Hospitalization is defined as initial hospitalization or prolongation of hospitalization for ≥ 24 hours, due to adverse event. | | | | | | | | | | | | |

11.1.2. Adverse events will be reported in accordance with the following guidelines:

11.1.3. Adverse event reports will be submitted in one of the following ways:

| (1) By email: (pdf) |
|---------------------|
| (2) By mail: |
| (3) By fax: |

<u>11.1.4.</u> An unexpected adverse event is defined as any adverse experience, the specificity or severity of which is not consistent with the risk information. This is a minimal risk study as both exercise and mobile app-driven interventions have been shown to improve outcomes in community-dwelling older adults.

11.1.5. A serious event refers to any event in which the outcome results in any of the following: death, a life-threatening adverse experience, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant disability, incapacity, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered a serious adverse drug experience when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition. We anticipate that any serious events will be related to standard of care cancer treatments and not due to the intervention. We will not collect adverse events related to cancer treatments.

<u>11.1.6.</u> Adverse events will be reported in accordance with institutional policies (University of Rochester, Research Subject Review Board, local IRB, URCC CCOP, CTO, and DSMB) as per their requirements.

#### 11.2. Data Safety Monitoring

- 11.2.1. All adverse events requiring reporting will be submitted to the current Project Coordinator as described in Section 11.1. Serious adverse event reports will be forwarded to the study chair and the Data Safety and Monitoring Committee (DSMC). Adverse events are entered into a protocol-specific spreadsheet.
- <u>11.2.2.</u> Adverse event rates are monitored utilizing the spreadsheet. If a serious adverse event is reported frequently, the study chair will conduct a detailed review. The DSMC Committee Chair will be notified and will determine if further action is required.
- 11.2.3. The Data Safety Monitoring Committee (DSMC) will review study progress and cumulative reports of adverse events every year and as needed. An overall assessment of accrual and adverse events will enable the committee members to assess whether significant benefits or risks are occurring that would warrant study closure.

#### 12.0 References

- 1. Ludmir EB, Mainwaring W, Lin TA, et al. Factors Associated With Age Disparities Among Cancer Clinical Trial Participants. *JAMA Oncol*. Jun 3 2019;doi:10.1001/jamaoncol.2019.2055
- 2. Burnett AK, Russell NH, Hills RK, et al. A comparison of clofarabine with ara-C, each in combination with daunorubicin as induction treatment in older patients with acute myeloid leukaemia. *Leukemia*. 2017//02/02 2017;31(2):310-317. doi:10.1038/leu.2016.225
- 3. Lancet JE, Uy GL, Cortes JE, et al. Final results of a phase III randomized trial of CPX-351 versus 7+3 in older patients with newly diagnosed high risk (secondary) AML. *Journal of Clinical Oncology*. 2016//05/05-20 2016;34(15\_suppl):7000-7000. doi:10.1200/JCO.2016.34.15 suppl.7000
- 4. Kantarjian HM, Thomas XG, Dmoszynska A, et al. Multicenter, randomized, open-label, phase III trial of decitabine versus patient choice, with physician advice, of either supportive care or low-dose cytarabine for the treatment of older patients with newly diagnosed acute myeloid leukemia. *Journal of Clinical Oncology: Official Journal of the American Society of Clinical Oncology*. 2012//07/07-20 2012;30(21):2670-2677. doi:10.1200/JCO.2011.38.9429
- 5. Juliusson G, Lazarevic V, Hörstedt A-S, Hagberg O, Höglund M. Acute myeloid leukemia in the real world: why population-based registries are needed. *Blood*. 2012//04/04-26 2012;119(17):3890-3899. doi:10.1182/blood-2011-12-379008
- 6. Khan C, Pathe N, Fazal S, Lister J, Rossetti JM. Azacitidine in the management of patients with myelodysplastic syndromes. *Ther Adv Hematol*. Dec 2012;3(6):355-73. doi:10.1177/2040620712464882
- 7. DiNardo CD, Pratz K, Pullarkat V, et al. Venetoclax combined with decitabine or azacitidine in treatment-naive, elderly patients with acute myeloid leukemia. *Blood*. Jan 3 2019;133(1):7-17. doi:10.1182/blood-2018-08-868752
- 8. Stein EM, DiNardo CD, Pollyea DA, et al. Enasidenib in mutant IDH2 relapsed or refractory acute myeloid leukemia. *Blood*. Aug 10 2017;130(6):722-731. doi:10.1182/blood-2017-04-779405
- 9. DiNardo CD, Pratz KW, Letai A, et al. Safety and preliminary efficacy of venetoclax with decitabine or azacitidine in elderly patients with previously untreated acute myeloid leukaemia: a non-randomised, open-label, phase 1b study. *Lancet Oncol*. Feb 2018;19(2):216-228. doi:10.1016/s1470-2045(18)30010-x
- 10. Shahrokni A, Loh KP, Wood WA. Toward Modernization of Geriatric Oncology by Digital Health Technologies. *Am Soc Clin Oncol Educ Book*. Mar 2020;40:1-7. doi:10.1200/edbk\_279505
- 11. Medeiros BC, Satram-Hoang S, Momin F, Parisi M. Real-World Treatment Patterns and Comparative Effectiveness Among a Population of Elderly Patients with Acute Myeloid Leukemia (AML). *Blood*. 2018;132(Supplement 1):835-835. doi:10.1182/blood-2018-99-111267
- 12. Klepin HD, Geiger AM, Tooze JA, et al. Geriatric assessment predicts survival for older adults receiving induction chemotherapy for acute myelogenous leukemia. *Blood*. 2013//05/05-23 2013;121(21):4287-4294. doi:10.1182/blood-2012-12-471680

- 13. Fallahzadeh R, Rokni SA, Ghasemzadeh H, Soto-Perez-de-Celis E, Shahrokni A. Digital Health for Geriatric Oncology. *JCO Clin Cancer Inform*. Dec 2018;2:1-12. doi:10.1200/cci.17.00133
- 14. Hoogland AI, Mansfield J, Lafranchise EA, Bulls HW, Johnstone PA, Jim HSL. eHealth literacy in older adults with cancer. *J Geriatr Oncol*. Jan 6 2020;doi:10.1016/j.jgo.2019.12.015
- 15. Poleshuck E, Wittink M, Crean H, et al. Using patient engagement in the design and rationale of a trial for women with depression in obstetrics and gynecology practices. *Contemporary clinical trials*. Apr 30 2015;43:83-92. doi:10.1016/j.cct.2015.04.010
- 16. Wittink MN, Cary M, Tenhave T, Baron J, Gallo JJ. Towards patient-centered care for depression: Conjoint methods to tailor treatment based on preferences. *Patient*. 2010;3(3):145-157. doi:10.2165/11530660
- 17. Eraker SA, Sox HC, Jr. Assessment of patients' preferences for therapeutic outcomes. *Medical decision making : an international journal of the Society for Medical Decision Making*. 1981;1(1):29-39.
- 18. O'Connor AM, Boyd NF, Tritchler DL, Kriukov Y, Sutherland H, Till JE. Eliciting preferences for alternative cancer drug treatments. The influence of framing, medium, and rater variables. *Medical decision making : an international journal of the Society for Medical Decision Making*. Winter 1985;5(4):453-63.
- 19. Hauber AB, Gonzalez JM, Groothuis-Oudshoorn CG, et al. Statistical Methods for the Analysis of Discrete Choice Experiments: A Report of the ISPOR Conjoint Analysis Good Research Practices Task Force. *Value Health*. Jun 2016;19(4):300-15. doi:10.1016/j.jval.2016.04.004
- 20. Wilson L, Loucks A, Bui C, et al. Patient centered decision making: use of conjoint analysis to determine risk-benefit trade-offs for preference sensitive treatment choices. *Journal of the neurological sciences*. Sep 15 2014;344(1-2):80-7. doi:10.1016/j.jns.2014.06.030
- 21. Loh KP, Xu H, Back A, et al. Patient-hematologist discordance in perceived chance of cure in hematologic malignancies: A multicenter study. *Cancer*. Dec 6 2019;doi:10.1002/cncr.32656
- 22. El-Jawahri A, Nelson-Lowe M, VanDusen H, et al. Patient-Clinician Discordance in Perceptions of Treatment Risks and Benefits in Older Patients with Acute Myeloid Leukemia. *Oncologist*. Feb 2019;24(2):247-254. doi:10.1634/theoncologist.2018-0317
- 23. Weeks JC, Cook EF, O'Day SJ, et al. Relationship between cancer patients' predictions of prognosis and their treatment preferences. *Jama*. Jun 3 1998;279(21):1709-14. doi:10.1001/jama.279.21.1709
- 24. Mack JW, Weeks JC, Wright AA, Block SD, Prigerson HG. End-of-life discussions, goal attainment, and distress at the end of life: predictors and outcomes of receipt of care consistent with preferences. *J Clin Oncol*. Mar 1 2010;28(7):1203-8. doi:10.1200/jco.2009.25.4672
- 25. Mack JW, Walling A, Dy S, et al. Patient beliefs that chemotherapy may be curative and care received at the end of life among patients with metastatic lung and colorectal cancer. *Cancer*. Jun 1 2015;121(11):1891-7. doi:10.1002/cncr.29250
- 26. Yennurajalingam S, Lu Z, Prado B, Williams JL, Lim KH, Bruera E. Association between Advanced Cancer Patients' Perception of Curability and Patients' Characteristics, Decisional

- Control Preferences, Symptoms, and End-of-Life Quality Care Outcomes. *J Palliat Med*. Jul 26 2018;doi:10.1089/jpm.2018.0186
- 27. Numico G, Anfossi M, Bertelli G, et al. The process of truth disclosure: an assessment of the results of information during the diagnostic phase in patients with cancer. *Annals of oncology: official journal of the European Society for Medical Oncology*. May 2009;20(5):941-5. doi:10.1093/annonc/mdn709
- 28. Brokalaki EI, Sotiropoulos GC, Tsaras K, Brokalaki H. Awareness of diagnosis, and information-seeking behavior of hospitalized cancer patients in Greece. *Support Care Cancer*. Nov 2005;13(11):938-42. doi:10.1007/s00520-005-0794-7
- 29. Caruso A, Di Francesco B, Pugliese P, Cinanni V, Corlito A. Information and awareness of diagnosis and progression of cancer in adult and elderly cancer patients. *Tumori*. May-Jun 2000;86(3):199-203.
- 30. Pinquart M, Sorensen S. Spouses, adult children, and children-in-law as caregivers of older adults: a meta-analytic comparison. *Psychol Aging*. Mar 2011;26(1):1-14. doi:10.1037/a0021863
- 31. Glajchen M. The emerging role and needs of family caregivers in cancer care. *J Support Oncol*. Mar-Apr 2004;2(2):145-55.
- 32. Dionne-Odom JN, Ejem D, Wells R, et al. How family caregivers of persons with advanced cancer assist with upstream healthcare decision-making: A qualitative study. *PLOS ONE*. 2019;14(3):e0212967. doi:10.1371/journal.pone.0212967
- 33. Wittenberg E, Borneman T, Koczywas M, Del Ferraro C, Ferrell B. Cancer Communication and Family Caregiver Quality of Life. *Behavioral sciences (Basel, Switzerland)*. Mar 2 2017;7(1)doi:10.3390/bs7010012
- 34. Waldron EA, Janke EA, Bechtel CF, Ramirez M, Cohen A. A systematic review of psychosocial interventions to improve cancer caregiver quality of life. *Psychooncology*. Jun 2013;22(6):1200-7. doi:10.1002/pon.3118
- 35. Wittenberg E, Buller H, Ferrell B, Koczywas M, Borneman T. Understanding Family Caregiver Communication to Provide Family-Centered Cancer Care. *Semin Oncol Nurs*. Dec 2017;33(5):507-516. doi:10.1016/j.soncn.2017.09.001
- 36. Zhang AY, Zyzanski SJ, Siminoff LA. Differential patient-caregiver opinions of treatment and care for advanced lung cancer patients. *Soc Sci Med*. Apr 2010;70(8):1155-8. doi:10.1016/j.socscimed.2009.12.023
- 37. Trevino KM, Prigerson HG, Shen MJ, et al. Association between advanced cancer patient-caregiver agreement regarding prognosis and hospice enrollment. *Cancer*. May 30 2019;doi:10.1002/cncr.32188
- 38. McPherson CJ, Wilson KG, Lobchuk MM, Brajtman S. Family caregivers' assessment of symptoms in patients with advanced cancer: concordance with patients and factors affecting accuracy. *J Pain Symptom Manage*. Jan 2008;35(1):70-82. doi:10.1016/j.jpainsymman.2007.02.038
- 39. Hsu T, Loscalzo M, Ramani R, et al. Are Disagreements in Caregiver and Patient Assessment of Patient Health Associated with Increased Caregiver Burden in Caregivers of Older Adults with Cancer? *Oncologist*. Nov 2017;22(11):1383-1391. doi:10.1634/theoncologist.2017-0085

- 40. Rodenbach RA, Norton SA, Wittink MN, et al. When chemotherapy fails: Emotionally charged experiences faced by family caregivers of patients with advanced cancer. *Patient Educ Couns*. May 2019;102(5):909-915. doi:10.1016/j.pec.2018.12.014
- 41. Sonnenblick M, Friedlander Y, Steinberg A. Dissociation between the wishes of terminally ill parents and decisions by their offspring. *J Am Geriatr Soc*. Jun 1993;41(6):599-604. doi:10.1111/j.1532-5415.1993.tb06729.x
- 42. Higginson IJ, Gao W. Caregiver assessment of patients with advanced cancer: concordance with patients, effect of burden and positivity. *Health Qual Life Outcomes*. Jun 2 2008;6:42. doi:10.1186/1477-7525-6-42
- 43. Loh KP, Abdallah M, Kadambi S, et al. Treatment decision-making in acute myeloid leukemia: a qualitative study of older adults and community oncologists. *Leuk Lymphoma*. Oct 11 2020:1-12. doi:10.1080/10428194.2020.1832662
- 44. Loh KP, Sanapala C, Digiovanni G, Mustian K, Klepin H, Janelsins M, Schnall R, Culakova E, Vertino P, Susiarjo M, Mendler J, Liesveld J, Mohile S. Qualitative study of a mobile health exercise intervention for older patients with myeloid neoplasms. Oral presentation at: University of Rochester Department Medicine Unmasked Conference; 27-29 May 2020, Rochester, New York, United States.
- 45. Acharya UH, Halpern AB, Wu QV, et al. Impact of region of diagnosis, ethnicity, age, and gender on survival in acute myeloid leukemia (AML). *J Drug Assess*. 2018;7(1):51-53. doi:10.1080/21556660.2018.1492925
- 46. Ostir GV, Volpato S, Fried LP, Chaves P, Guralnik JM. Reliability and sensitivity to change assessed for a summary measure of lower body function: results from the Women's Health and Aging Study. *J Clin Epidemiol*. Sep 2002;55(9):916-21. doi:10.1016/s0895-4356(02)00436-5
- 47. Marsh AP, Wrights AP, Haakonssen EH, et al. The Virtual Short Physical Performance Battery. *J Gerontol A Biol Sci Med Sci*. 2015;70(10):1233-1241. doi:10.1093/gerona/glv029
- 48. Shelkey M, Wallace M. Katz Index of Independence in Activities of Daily Living. *Home Healthcare Now*. 2001;19(5)
- 49. Graf C. The Lawton instrumental activities of daily living scale. *The American journal of nursing*. Apr 2008;108(4):52-62; quiz 62-3. doi:10.1097/01.Naj.0000314810.46029.74
- 50. Hurria A, Togawa K, Mohile SG, et al. Predicting chemotherapy toxicity in older adults with cancer: a prospective multicenter study. *Journal of clinical oncology : official journal of the American Society of Clinical Oncology*. 2011;29(25):3457-3465. doi:10.1200/JCO.2011.34.7625
- 51. Fillenbaum GG, Smyer MA. The development, validity, and reliability of the OARS multidimensional functional assessment questionnaire. *J Gerontol*. Jul 1981;36(4):428-34. doi:10.1093/geronj/36.4.428
- 52. Löwe B, Decker O, Müller S, et al. Validation and standardization of the Generalized Anxiety Disorder Screener (GAD-7) in the general population. *Medical care*. Mar 2008;46(3):266-74. doi:10.1097/MLR.0b013e318160d093
- 53. Durmaz B, Soysal P, Ellidokuz H, Isik AT. Validity and reliability of geriatric depression scale-15 (short form) in Turkish older adults. *North Clin Istanb*. 2018;5(3):216-220. doi:10.14744/nci.2017.85047
- 54. Kroenke K, Spitzer RL, Williams JB. The Patient Health Questionnaire-2: validity of a two-item depression screener. *Med Care*. Nov 2003;41(11):1284-92. doi:10.1097/01.Mlr.0000093487.78664.3c

- 55. Fillenbaum GG. Multidimensional functional assessment of older adults: the Duke Older Americans Resources and Services procedures / Gerda G. Fillenbaum. L. Erlbaum Associates; 1988.
- 56. Borson S, Scanlan J, Brush M, Vitaliano P, Dokmak A. The mini-cog: a cognitive 'vital signs' measure for dementia screening in multi-lingual elderly. *International journal of geriatric psychiatry*. Nov 2000;15(11):1021-7. doi:10.1002/1099-1166(200011)15:11<1021::aid-gps234>3.0.co;2-6
- 57. Maly RC, Frank JC, Marshall GN, DiMatteo MR, Reuben DB. Perceived efficacy in patient-physician interactions (PEPPI): validation of an instrument in older persons. *Journal of the American Geriatrics Society*. Jul 1998;46(7):889-94. doi:10.1111/j.1532-5415.1998.tb02725.x
- 58. Moore CD, Cook KM. Promoting and measuring family caregiver self-efficacy in caregiver-physician interactions. *Soc Work Health Care*. 2011;50(10):801-14. doi:10.1080/00981389.2011.580835
- 59. Reeve BB, Thissen DM, Bann CM, et al. Psychometric evaluation and design of patient-centered communication measures for cancer care settings. *Patient Educ Couns*. Jul 2017;100(7):1322-1328. doi:10.1016/j.pec.2017.02.011
- 60. Kriston L, Scholl I, Hölzel L, Simon D, Loh A, Härter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. *Patient Education and Counseling*. 2010/07/01/ 2010;80(1):94-99. doi:https://doi.org/10.1016/j.pec.2009.09.034
- 61. Calderon C, Ferrando PJ, Carmona-Bayonas A, et al. Validation of SDM-Q-Doc Questionnaire to measure shared decision-making physician's perspective in oncology practice. *Clin Transl Oncol*. Nov 2017;19(11):1312-1319. doi:10.1007/s12094-017-1671-9
- 62. Forcino RC, Barr PJ, O'Malley AJ, et al. Using CollaboRATE, a brief patient-reported measure of shared decision making: Results from three clinical settings in the United States. *Health Expect*. Feb 2018;21(1):82-89. doi:10.1111/hex.12588
- 63. Bennett C, Graham ID, Kristjansson E, Kearing SA, Clay KF, O'Connor AM. Validation of a preparation for decision making scale. *Patient Educ Couns*. Jan 2010;78(1):130-3. doi:10.1016/j.pec.2009.05.012
- 64. Degner LF, Sloan JA, Venkatesh P. The Control Preferences Scale. *Can J Nurs Res*. Fall 1997;29(3):21-43.
- 65. O'Connor AM. Validation of a decisional conflict scale. *Med Decis Making*. Jan-Mar 1995;15(1):25-30. doi:10.1177/0272989x9501500105
- 66. Brehaut JC, O'Connor AM, Wood TJ, et al. Validation of a decision regret scale. *Med Decis Making*. Jul-Aug 2003;23(4):281-92. doi:10.1177/0272989x03256005
- 67. Rost L, Chen Y, Fain RS, 3rd, et al. "Was It Worth It?": A Pilot Study in Patient Perspectives on the Worthwhileness of Radiation Therapy. *Am J Clin Oncol*. Aug 2020;43(8):598-601. doi:10.1097/coc.000000000000011
- 68. Grochtdreis T, Dams J, König HH, Konnopka A. Health-related quality of life measured with the EQ-5D-5L: estimation of normative index values based on a representative German population sample and value set. *Eur J Health Econ*. Aug 2019;20(6):933-944. doi:10.1007/s10198-019-01054-1

- 69. Peres S, Pham T, Phillips R. Validation of the System Usability Scale (SUS). *Proceedings of the Human Factors and Ergonomics Society Annual Meeting*. 09/30 2013;57:192-196. doi:10.1177/1541931213571043
- 70. Ryff CD. Happiness is everything, or is it? Explorations on the meaning of psychological well-being. *Journal of Personality and Social Psychology*. 1989;57(6):1069-1081. doi:10.1037/0022-3514.57.6.1069
- 71. Little R, Yau L. Intent-to-treat analysis for longitudinal studies with drop-outs. *Biometrics*. Dec 1996;52(4):1324-33.
- 72. Hsieh HF, Shannon SE. Three approaches to qualitative content analysis. *Qual Health Res.* Nov 2005;15(9):1277-88. doi:10.1177/1049732305276687
- 73. Loh KP, Ramsdale E, Culakova E, et al. Novel mHealth App to Deliver Geriatric Assessment-Driven Interventions for Older Adults With Cancer: Pilot Feasibility and Usability Study. *JMIR Cancer*. Oct 29 2018;4(2):e10296. doi:10.2196/10296
- 74. Nielsen J, Landauer TK. A mathematical model of the finding of usability problems. CHI '93 Conference on Human Factors in Computing Systems; 1993; Amsterdam, The Netherlands. 1993. Pp. 206–213.
- 75. Virzi RA. Refining the Test Phase of Usability Evaluation: How Many Subjects Is Enough? *Human Factors*. 1992/08/01 1992;34(4):457-468. doi:10.1177/001872089203400407
- 76. Fraenkel L. Feasibility of Using Modified Adaptive Conjoint Analysis Importance Questions. *Patient*. 2010;3(4):209-215. doi:10.2165/11318820-000000000-00000
- 77. Dwight-Johnson M, Lagomasino IT, Aisenberg E, Hay J. Using conjoint analysis to assess depression treatment preferences among low-income Latinos. *Psychiatr Serv*. Aug 2004;55(8):934-6. doi:10.1176/appi.ps.55.8.934
- 78. Clayman ML, Makoul G, Harper MM, Koby DG, Williams AR. Development of a shared decision making coding system for analysis of patient-healthcare provider encounters. *Patient Educ Couns*. Sep 2012;88(3):367-72. doi:10.1016/j.pec.2012.06.011
- 79. Elwyn G, Edwards A, Wensing M, Hood K, Atwell C, Grol R. Shared decision making: developing the OPTION scale for measuring patient involvement. *Qual Saf Health Care*. Apr 2003;12(2):93-9. doi:10.1136/qhc.12.2.93
- 80. Harris PA, Taylor R, Thielke R, Payne J, Gonzalez N, Conde JG. Research electronic data capture (REDCap)--a metadata-driven methodology and workflow process for providing translational research informatics support. *J Biomed Inform*. Apr 2009;42(2):377-81. doi:10.1016/j.jbi.2008.08.010
- 81. Clinical & Translational Science Institute. REDCap. REDCap at the University of Rochester. Available at: <a href="https://www.urmc.rochester.edu/ctsi/research-help/REDCap.cfm">https://www.urmc.rochester.edu/ctsi/research-help/REDCap.cfm</a>.